CLINICAL TRIAL: NCT01891773
Title: Improving Pediatric Asthma Care Through Inhaled Steroids in Schools (ISIS)
Brief Title: Improving Pediatric Asthma Care Through Inhaled Steroids in Schools
Acronym: ISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Stephen J. Teach, MD, MPH, Associate Chief, Division of Emergency Medicine, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00003859
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
Keywords: Asthma; Inhaled Corticosteroids; School Nurses
MeSH Terms: conditions — Asthma | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- School-based therapy (Experimental): Daily dose of medication to be provided in the school setting.
  Interventions: Behavioral: Inhaled steroids in school.
- Usual Care (No Intervention): Daily medication to be taken at home.

INTERVENTIONS:
Behavioral: Inhaled steroids in school. — Morning dose of inhaled steroids given in school by school nurse instead of at home.
  Arms: School-based therapy

SUMMARY:
Asthma is the most common chronic pediatric disease in the United States, and is the most common cause of school absenteeism due to a chronic disease. Socioeconomically disadvantaged minority children receive disproportionately poor asthma care and incur a disproportionate share of asthma-related morbidity. The District of Columbia is particularly severely affected, with a lifetime asthma prevalence rate among children 0-17 years of age in 2010 of 22%, more than double the national average.

One of the major challenges in treating asthma is poor adherence to daily controller medications, particularly inhaled corticosteroids (ICS) which are the cornerstone of the NIH guidelines for asthma management. In an attempt to overcome poor compliance, investigators in Rochester, New York have partnered with primary care providers in their community to arrange for ICS administration at school by school nurses, and this approach yielded significant improvements in several asthma outcomes.

The investigators propose to collaborate in a pilot research project with the overall goal of improving asthma outcomes through reducing barriers to medication adherence. Specifically, the investigators aim to improve adherence to controller medications (inhaled corticosteroids - ICS) among DC children with asthma through the following activities:

1. A pilot prospective randomized clinical trial of home vs. school administration of ICS among DC children in grades kindergarten-8 with persistent asthma.
2. Qualitative interviews with nurses from DC public and public charter school to identify key barriers to administration of daily controller medications in the school setting

ELIGIBILITY:
Inclusion Criteria:

* Current enrollment in one of the grades K-8 at a DC public school (DCPS) or DC public charter school (DCPCS)
* Active public insurance
* Persistent asthma
* An Asthma Action Plan including daily ICS
* Child's primary asthma caregiver present, meaning the person who usually takes care of his/her asthma at home and can answer questions about his/her medical history.

Exclusion Criteria:

* Chronic disease of the cardio-pulmonary system other than asthma
* Non-English speaking parent/guardian
* Currently enrolled in in another asthma study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion of doses received | 60 day treatment period
  Proportion of doses of ICS received during the 60 days outcome period

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Teach, MD, MPH, Principal Investigator — Children's National Research Institute